CLINICAL TRIAL: NCT02998359
Title: Randomised Controlled Trial of Hemiarthroplasty Versus Total Hip Replacement for Intracapsular Hip Fractures
Brief Title: Hemiarthroplasty Versus Total Hip Replacement for Intracapsular Hip Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peterborough and Stamford Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Martyn J Parker, Consultant orthopaedic surgeon, Peterborough and Stamford Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R&D/2012/30
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2018-04

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Hemiarthroplasty; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemiarthroplasty (Active Comparator): A cemented polished double taper stem hemiarthroplasty inserted via an anterior-lateral surgical approach (Zimmer incorporated, UK).
  Interventions: Device: Hemiarthroplasty
- Total hip replacment (Active Comparator): A cemented polished double taper stem arthroplasty inserted via an anterior-lateral surgical approach with a cemented acetabular cup (Zimmer incorporated, UK).
  Interventions: Device: Total hip arthroplasty

INTERVENTIONS:
Device: Hemiarthroplasty — A cemented polished double taper stem hemiarthroplasty inserted via an anterior-lateral surgical approach (Zimmer incorporated, UK).
  Arms: Hemiarthroplasty
Device: Total hip arthroplasty — A cemented polished double taper stem arthroplasty stem inserted via an anterior-lateral surgical approach with a cemented acetabular cup (Zimmer incorporated, UK).
  Arms: Total hip replacment

SUMMARY:
In England each year over 9,000 people fracture their hip. Most of these are elderly females with the fracture occurring after a fall. Approximately half of these fractures are classified as intracapsular fractures because of their close proximity to the hip joint. The majority of these fractures are treated surgically by excising the broken femoral neck and removing the femoral head (ball part of the hip joint) and replacing it with an artificial hip joint. This hip replacement has traditionally been a hemiarthroplasty or sometimes termed a 'half hip replacement' in which only the ball part of the hip joint is replaced.

An alternative type of hip replacement is the full total hip replacement in which the socket part of the joint is also replaced. This is the operation that is used for replacing arthritic hips. In recent years there have been a number of randomised trials that have compared the outcome for patients with an intracapsular hip fracture treated with either a partial hip replacement (hemiarthroplasty) against those treated with a total hip replacement (THR). Results to date have suggested slightly better long term functional results for those treated with a THR, but it still remains unclear if these benefits are offset by the increased surgical complexity of the procedure and the extra cost involved for a THR.

At present the numbers of studies on this topic are too few with limited patient numbers to make any definite conclusions. This study aims to add to the research studies by comparing the two surgical procedures, to enable orthopaedic surgeons to determine the optimum surgical treatment for this common and disabling condition.

DETAILED DESCRIPTION:
The trial will be run as close to the ideal trial methodology for a randomised trial as specified by the CONSORT statement as possible. This will include secure randomisation, intention to treat analysis, full reporting of outcomes and follow-up by a person who is blinded to the prosthesis used. The trial will follow the code of good clinical practice as specified by the hospital trusts Research and Development Committee.

In Peterborough all hip fracture patients are admitted to the acute trauma ward and transferred to the care of MJP. Those patients that are willing to participant in one of our randomised trials are consented prior to surgery. Treatment follows standard evidence based protocols with follow-up of all patients in a hip fracture clinic. A comprehensive database is maintained for all patients containing both audit and research data. Included in this is a standardised assessment of outcome.

The surgical treatments under comparison will be either a cemented Exeter stem monoblock prosthesis inserted via an anteriolateral surgical approach or a cemented Total hip replacement. The stem for the THR will be a polished tapered stem of the Exeter type with a 32 or 36mm head articulating with a cemented high density polyethylene cemented acetabular cup. All operations will be undertaken or supervised by MJP. Post-operative care programmes for the two patients will be identical.

After discharge patient will be seen once in the hip fracture clinic by MJP. At this time they will also be assessed by the research nurse who is blinded to the type of prosthesis used. The outcome questionnaire is completed which includes an assessment of hip movement and limb shortening. All subsequent follow-up assessments will be done by phone call from the research nurse. Any patient with significant residual symptoms will be asked to re-attend the hip fracture clinic.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Peterborough District Hospital with a displaced intracapsular fracture will be considered for inclusion in the study. Patients will need to be

  * able to walk independently out of doors with no more than the use of a stick
  * not cognitively impaired
  * medically fit for anaesthesia for either procedure

Exclusion Criteria:

* • Those aged less than 50 years (these patient have an expected good long term survival and are all treated by reduction and internal fixation).

  * All other patients in which the injury is to be treated by reduction and internal fixation.
  * Those with impaired mobility prior to the injury (defined as not able to walk out of doors with no more than the use of a stick).
  * Patients who are not considered to be medically fit for either procedure.
  * Patients who decline to participate.
  * Patients with senile dementia and those without the capacity to give informed consent. These patients are defined as those with a standard mental test score of lower than 5 our of 10. (These patients from previous studies have been found to be at increased risk of dislocation and post-operative complications after THR and this method of treatment is not recommended for this group).
  * Patients admitted when MJP is not available to supervise treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change in a mobility score | at one year from injury
  A nine point mobility score - Parker MJ, Palmer CR. A new mobility score for predicting mortality after hip fracture. J Bone Joint Surg 1993;75-B:797-8.

CONTACTS AND LOCATIONS:
Locations (1):
- Peterborough City Hospital, Peterborough, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
not IPD anticipated

REFERENCES:
- [Result] Parker MJ, Cawley S. Treatment of the displaced intracapsular fracture for the 'fitter' elderly patients: A randomised trial of total hip arthroplasty versus hemiarthroplasty for 105 patients. Injury. 2019 Nov;50(11):2009-2013. doi: 10.1016/j.injury.2019.09.018. Epub 2019 Sep 10. PMID 31543318